CLINICAL TRIAL: NCT03049696
Title: An Integrated Surgical and Physical Activity Program to Identify Bariatric Surgery Quality Indicators and Evaluate Patient Outcomes and Quality of Life
Brief Title: Does Participation in a Pre-Operative Physical Activity Program Improve Patient Outcomes and Quality of Life?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Victoria General Hospital Foundation (Unknown)
Responsible Party: Principal Investigator, Dr. Krista Hardy, Co-Principal Investigator, University of Manitoba
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2016:283
Record Dates: First submitted 2017-01-18; First posted 2017-02-10 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Obesity; Bariatric Surgery; Roux-En-Y Gastric Bypass; Exercise; Quality of Life
Keywords: Roux-En-Y Gastric Bypass; Bariatric Surgery; Pre-Operative Physical Activity and Education Program; Obesity; Exercise; Behaviour Modification; Surgical Outcomes; Quality of Life
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Control Group: Publically funded bariatric surgery program administered through the Centre for Bariatric and Metabolic Surgery (CMBS).; Matched control group Intervention Group: CMBS Program standard of care plus the ENCOURAGING START Program (University of Manitoba Active Living Centre)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Standard of Care) (No Intervention): All patients will receive the Centre for Metabolic and Bariatric Surgery (CMBS) standard of care including two to four multidisciplinary visits over six months, exercise counseling (kinesiologist), completion of a the CMBS behavior modification program (Craving ChangeTM), and achievement of lifestyle and dietary modification goals in order to be scheduled for surgery. The standard of care will be used as the control group (n=24). Matched historical controls (1:1) will be selected (based on age, gender, and body mass index) from the existing CMBS database.
- Intervention Group-ENCOURAGEING START (Experimental): Intervention group participants (n=24) will receive the standard of care and complete a 16-week supervised physical activity/behaviour modification program at no cost. The first eight weeks of the program involves structured exercise (two per week) and education classes that patients must attend. Progression to a moderate/high-intensity interval program based the patient's capabilities will occur. Participants will also attend education sessions on risk factor reduction, healthy eating, exercise, stress management and promotion of self-managed care. During the second eight week period, participants will be given access to attend drop-in exercise classes or can opt to complete at home exercise. Participants will have an opportunity to meet with the kinesiologist on at least 4 occasions (60 minutes/meeting) for additional physical activity counseling and assistance with overcoming barriers preventing physical activity.
  Interventions: Behavioral: ENCOURAGEING START

INTERVENTIONS:
Behavioral: ENCOURAGEING START — 16-week physical activity and behaviour modification/education program. CMBS approved bariatric surgery patients participate in structured, supervised physical activity sessions (2 per week) and behaviour modification-education classes during weeks 1 through 8. During weeks 9 through 16, patients will be given access to attend drop in physical activity sessions or can opt to complete physical activity at home.
  Other Names: Physical activity and behaviour modification/education program
  Arms: Intervention Group-ENCOURAGEING START

SUMMARY:
The primary objective of the study is to determine whether participation in a pre-bariatric surgery physical activity and behavior modification/education program (ENCOURAGEING START) that is tailored to the unique needs of obese bariatric surgery patients, improves physical fitness, surgical outcomes, patient health and quality of life. Short- (one year) and long- (five year) term outcomes will be compared to matched historical controls (1:1) based on age, gender, and body mass index (BMI) from the existing Manitoba Centre for Metabolic and Bariatric Surgery (CMBS) database. Our findings will determine whether a pre-bariatric surgery physical activity and behavior modification/education program results in improve surgical and patient outcomes and inform the development of evidence-based physical activity (PA) guidelines for bariatric surgery patients and improved CMBS program delivery.

DETAILED DESCRIPTION:
The objective of this study is to design and implement a 16-week pre-operative physical activity and behaviour modification/education program (ENCOURAGEING Start) based on a collaborative partnership among the Centre for Metabolic and Bariatric Surgery (CMBS), the University of Manitoba Faculty of Kinesiology and Recreation Management, and Victoria General Hospital (VGH). Twenty-four CMBS patients, approved for bariatric surgery, will participate in the 16 week ENCOURAGEING START program. The goal is to develop evidence-based pre-operative physical activity (PA) guidelines and tools to improve bariatric surgery program delivery and patient outcomes. All patients will receive the Centre for Metabolic and Bariatric Surgery (CMBS) standard of care including two to four multidisciplinary visits over six months, exercise counseling from a kinesiologist, completion of a behavior modification program (Craving ChangeTM), and achievement of lifestyle and dietary modification goals in order to be scheduled for surgery. An interdisciplinary team of nurses, psychologists, dietitians, kinesiologists, anesthetists and internal medicine professionals participate in patient preparation. Intervention group participants will also complete the 16-week supervised physical activity and behaviour modification/education program (ENCOURAGEING START) at no cost. The first eight weeks of the ENCOURAGEING START program is a structured exercise and education period that patients must attend. During the second eight week period, opportunities for drop-in physical activity will be provided or patients can opt for at home exercise. Patient participation in physical activity will be monitored and follow-up with their experiences will be completed (by phone/email). A successfully developed and tested evidence-based physical activity promotion model (designed by co-applicant Dr. Todd Duhamel) has been tailored to the unique needs of the bariatric surgery patient population. It has been been shown successful at increasing weekly physical activity levels in patients with Body Mass Indexes (BMIs) between 30 to 35 and targets the physical and psycho-social-cognitive aspects of health. The intervention will be delivered by a kinesiologist (Certified Exercise Physiologist). Intervention group participants will complete two sessions of supervised, structured exercise classes per week for eight weeks. Progression to a moderate/high-intensity interval program based the patient's capabilities will occur. This approach has been shown to be safe and effective in the bariatric patient population. Participants will also attend education sessions on risk factor reduction, healthy eating, physical activity/exercise, stress management and promotion of self-managed care. Principles of shared decision-making will be utilized so providers and patients involved in the intervention will have shared control of treatment decisions. During the second eight week interval of the 16-week intervention, participants will be provided with access to facilitate attendance at drop-in exercise classes at the Active Living Centre (University of Manitoba). Participants will have the opportunity to meet with the kinesiologist on at least four occasions (60 minutes per meeting) throughout the 16-week intervention. This will provide participants with additional physical activity counseling if they would like more support to overcome the barriers that have prevented them from being physically active in the past. This counseling (and referral aspect) of the model builds upon the earlier experiences in the program and recognizes the importance of support from colleagues, friends and family. Participant attendance during the 16-week intervention will be monitored. In order to ensure adequate participation rates for this study, participant follow-up will be completed by telephone or email (based on participant consent and preference). All patients complete a liquid diet (900 calories per day) for two weeks prior to their surgery in order to reduce intra-abdominal obesity and facilitate the procedure. The study will follow the intension to treat (ITT) model and patient exclusion/withdrawal will be documented and reported according to the CONSORT guidelines. A time series quasi-experimental design will be used to document changes in outcome measures. Short (one year) and long-term (five year) outcomes will be compared to matched historical controls 1:1 based on age, gender, BMI from the existing CMBS database with the goal to determine whether participation in the program improves physical fitness, surgical outcomes, patient health and quality of life for obese patients. The primary outcome of the study is the change in the 6-minute walk test (6MWT) that measures the distance a patient walks in six minutes, unassisted and at a self-selected pace; a validated measure of physical fitness and a well-established measure of functional capacity that is easily tested and in expensive to administer. The 6MWT has been used to measure improvements in functional capacity in pre- and post-bariatric surgery studies. The secondary outcomes include anthropometric measurements (height and weight, BMI (kg/m2), neck circumference, waist and hip circumference, and body composition (Bioelectric Impedance Analysis; BIA), strength measurements (sit to stand and half-squat tests to assess dynamic balance, flexibility and muscular endurance, and the hand grip and arm curl tests to assess upper limb muscle strength and dynamic muscular endurance of the biceps), physical activity level (Actigraph accelerometer), cardiovascular disease risk measurement (blood pressure, total, LDL, and HDL cholesterol and triacylglyceride measurements, blood glucose, HA1c, small and large artery elasticity), frailty measurement, patient quality of life/satisfaction/mental health and depression surveys (Laval Health Related Quality of Life Questionnaire, PHQ9 and HAM-D; see included surveys), Self-compassion, anxiety and physical activity questionnaires, and CMBS program outcome measures (surgical complication rate, hospital length of stay, comorbidity resolution, continued participation in physical activity, weight loss, and weight loss maintenance). Tests at Week 0 (pre-intervention) include the 6MWT, anthropometric, body composition, strength, physical activity level (accelerometer), quality of life/mental health surveys, cardiovascular/ diabetes disease risk measurement, frailty measurement, and arterial elasticity. Tests at week 16 (post-intervention) and 12 months (post-operative) will include 6MWT, anthropometric, strength, physical activity level (accelerometer), quality of life/mental health patient satisfaction surveys, cardiovascular/ diabetes disease risk measurement, frailty measurement, and arterial elasticity. The quality of life/mental health patient satisfaction surveys will be also be completed at the 5 years post-operative period. Two REDCap databases (Data and Survey) will be designed and implemented to facilitate data collection of surgical and patient outcomes, longitudinal survey deployment and patient responses. The surgical outcome metrics are based on the American Society for Metabolic and Bariatric Surgery's (ASMBS) quality indicators for bariatric surgery with the goal to inform and define standardized outcome measures for RYGB surgery in Manitoba and Canada.

ELIGIBILITY:
Inclusion Criteria:

* Male and female obese adults (Body Mass Index equal to or greater than 35 and under 55);
* over 18 years old,
* approved for publicly funded Roux-en-Y gastric bypass surgery by the Centre for Metabolic and Bariatric Surgery,
* able to attend the regular training and education sessions of the intervention program.

Exclusion Criteria:

* Exclusion criteria include any orthopedic, neurologic or cardiopulmonary conditions that preclude moderately strenuous exercise,
* Body Mass Index over 55 (super-obese),
* sleeve gastrectomy, and
* the inability to commit to attending the regular training and education sessions of the intervention program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Six Minute Walk Test (6MWT) | Baseline (0 weeks), 8 weeks, 16 weeks, one year.
  Measures the distance a patient walks, unassisted and at a self-selected pace, in six minutes. A validated measure of physical fitness and a well-established measure of functional capacity. Has been used to measure improvements in functional capacity in pre- and post- bariatric surgery patients.

SECONDARY OUTCOMES:
Anthropometric Measurements-1 | Baseline (0 weeks), 8 weeks, 16 weeks, one and five years.
  Height (cm)
Anthropometric Measurements-2 | Baseline (0 weeks), 8 weeks, 16 weeks, one and five years.
  Body Mass Index (kg/m2)
Anthropometric Measurements-3 | Baseline (0 weeks), 8 weeks, 16 weeks, one and five years.
  Neck circumference (cm)
Anthropometric Measurements-4 | Baseline (0 weeks), 8 weeks, 16 weeks, one and five years.
  Waist circumference (cm)
Anthropometric Measurements-5 | Baseline (0 weeks), 8 weeks, 16 weeks, one and five years.
  Hip circumference (cm)
Anthropometric Measurements-6 | Baseline (0 weeks), 8 weeks, 16 weeks, and one year.
  Body composition (Bioelectric Impedance Analysis)
Anthropometric Measurements-7 | Baseline (0 weeks), 8 weeks, 16 weeks, one and five years.
  Weight (kg)
Strength Measurements-1 | Baseline (0 weeks), 8 weeks,16 weeks, and one year
  Half-squat test (to assess dynamic balance, flexibility and muscular endurance).
Strength Measurements-2 | Baseline (0 weeks), 8 weeks,16 weeks, and one year
  Hand grip test (to assess upper limb muscle strength and dynamic muscle endurance of the biceps).
Strength Measurements-3 | Baseline (0 weeks), 8 weeks,16 weeks, and one year
  Sit to stand test (to assess dynamic balance, flexibility and muscular endurance).
Strength Measurements-4 | Baseline (0 weeks), 8 weeks,16 weeks, and one year
  Arm curl tests (to assess upper limb muscle strength and dynamic muscle endurance of the biceps).
Physical Activity Level | Baseline (0 weeks), 8 and 16 weeks; one year.
  Measured using the Actigraph accelerometer. Each patient will be issued an Actigraph accelerometer that will track their physical activity level.
Cardiovascular Disease Risk Measurement-1 | Baseline (0 weeks), 8 weeks, 16 weeks and one year.
  Blood pressure (mmHg)
Cardiovascular Disease Risk Measurement-2 | Baseline (0 weeks), 16 weeks and one year.
  Total cholesterol
Cardiovascular Disease Risk Measurement-3 | Baseline (0 weeks), 16 weeks and one year.
  LDL cholesterol
Cardiovascular Disease Risk Measurement-4 | Baseline (0 weeks), 16 weeks and one year.
  HDL cholesterol
Cardiovascular Disease Risk Measurement-5 | Baseline (0 weeks), 16 weeks and one year.
  Blood triacylglyceride measurement
Cardiovascular Disease Risk Measurement-6 | Baseline (0 weeks), 16 weeks and one year.
  Blood glucose
Cardiovascular Disease Risk Measurement-7 | Baseline (0 weeks), 16 weeks and one year.
  Blood glycosylated hemoglobin (HA1c)
Cardiovascular Disease Risk Measurement-8 | Baseline (0 weeks), 8 weeks, 16 weeks and one year.
  Small artery elasticity
Cardiovascular Disease Risk Measurement-9 | Baseline (0 weeks), 8 weeks, 16 weeks and one year.
  Large artery elasticity.
Patient quality of life, satisfaction, and mental health-1 | Baseline (0 weeks), 8 weeks, 16 weeks; one and five years.
  Laval Health Related Quality of Life Questionnaire.
Patient quality of life, satisfaction, and mental health-2 | Baseline (0 weeks), 8 weeks, 16 weeks; one and five years.
  Patient Satisfaction Questionnaire (PSQ-18)
Patient quality of life, satisfaction, and mental health-3 | Baseline (0 weeks), 8 weeks, 16 weeks; one and five years.
  Patient Health Questionnaire (PHQ-9)
Self-Compassion, Anxiety, and Physical Activity Questionnaires | Baseline (0 weeks), 8 weeks, 16 weeks; one and five years.
  Various surveys assembled into one questionnaire package; Self-Compassion Scale, multi-dimensional Health Questionnaire (MHQ)-Health Anxiety Sub-Scale, Affective Responses to a Real Health Problem, Response to Illness Questionnaire, Physical Activity Intentions, Social Physique Anxiety Scale, Body Appreciation Scale-2, Exercise Task Self-Efficacy, and Exercise Regulations Questionnaire (BREQ-3).
Patient quality of life, satisfaction, and mental health-4 | Baseline (0 weeks), 8 weeks, 16 weeks; one and five years.
  Hospital Anxiety and Depression Scale (HADS),
Surgical Outcome Measures-1 | one year
  Surgical complication rate.
Surgical Outcome Measures-2 | one year
  Hospital length of stay.
Surgical Outcome Measures-3 | one year
  Comorbidity resolution.
Surgical Outcome Measures-4 | one year
  Continued participation in physical activity.
Surgical Outcome Measures-5 | one year
  Weight loss (amount; kg).
Surgical Outcome Measures-6 | one year
  Weight loss maintenance.

CONTACTS AND LOCATIONS:
Overall Officials: Krista M Hardy, MD, MSC, FRCSC, FACS, Principal Investigator — University of Manitoba
Locations (1):
- Centre for Metabolic and Bariatric Surgery (CMBS), Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.